CLINICAL TRIAL: NCT01060527
Title: Altered Faecal Protease Activity in Irritable Bowel Syndrome Patients in China
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: the second affiliated hospital of xi'an jiaotong university, the second affiliated hospital of xi'an jiaotong university
Other Study IDs: xi'an JTU091202
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome,protease activity,China
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (3):
- IBS-D
- IBS-C
- Controll

SUMMARY:
Irritable bowel syndrome (IBS) is a functional gastrointestinal disorder haracterised by abdominal pain or discomfort associated with altered bowel habits,while the mechanism is still not understood.Recent advances have conceptualized the faecal supernatants of diarrhoea-predominant IBS have a substantially higher serine protease activity, while in china,almost no studies have reported about protease activity in IBS.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the Rome III criteria for IBS participated in the study -

Exclusion Criteria:

* Organic gastrointestinal disorders were excluded by detailed blood and stool analyses, serological assays and colonoscopy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients in the second affiliated hospital of xi'an jiaotong university
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-01